CLINICAL TRIAL: NCT02764762
Title: An Open-Label, Phase 4 Study to Evaluate the Efficacy and Safety of Triple Combination Therapy With Vedolizumab IV, Adalimumab SC, and Oral Methotrexate in Early Treatment of Subjects With Crohn's Disease Stratified at Higher Risk for Developing Complications
Brief Title: Triple Combination Therapy in High Risk Crohn's Disease (CD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-4006; U1111-1175-9094 (Registry Identifier: WHO)
Record Dates: First submitted 2016-05-05; First posted 2016-05-06 (Estimated); Results first posted 2021-10-21 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab; Adalimumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral) (Experimental): In Triple Combination Therapy Phase, vedolizumab 300 mg, intravenous (IV) infusion, once at Weeks 0, 2, 6, 14 and 22, with adalimumab 160 mg subcutaneously (SC), once at Week 0, then 80 mg once at Week 2, then 40 mg once at Week 4 and every 2 weeks thereafter until Week 26 along with oral methotrexate 15 mg tablets orally once weekly from Weeks 0 up to Week 34. In Monotherapy Phase, vedolizumab 300 mg IV infusion once at Weeks 30, 38, 46, 54, 62, 70, 78, 86, 94 and 102.
  Interventions: Drug: Vedolizumab; Drug: Adalimumab; Drug: Methotrexate

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab intravenous infusion.
  Other Names: Entyvio; MLN0002 IV
Drug: Adalimumab — Adalimumab injection for subcutaneous use.
  Other Names: Humira
Drug: Methotrexate — Methotrexate oral tablets.

SUMMARY:
The purpose of this study is to determine the effect of triple combination therapy with an anti-integrin (vedolizumab intravenous [IV]), a tumor necrosis factor (TNF) antagonist (adalimumab subcutaneously [SC]), and an immunomodulator (oral methotrexate) on endoscopic remission in participants with newly-diagnosed CD stratified at higher risk for complications.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat people who have CD. This study will look at the endoscopic remission and mucosal healing of gastrointestinal tract of people who take vedolizumab as triple combination therapy with adalimumab and methotrexate.

The study will enroll approximately 60 participants. Participants will receive triple combination therapy which includes:

* Vedolizumab 300 mg (intravenous)
* Adalimumab 160/80/40 mg (subcutaneous)
* Methotrexate 15 mg (oral)

All participants will receive vedolizumab intravenous infusion on Weeks 0, 2, 6, 14 and 22 along with adalimumab 160 mg, subcutaneous injection at Week 0, 80 mg at Week 2, then 40 mg once at Week 4 and every 2 weeks thereafter until Week 26 along with methotrexate tablets orally, once weekly from Weeks 0 up to Week 34. In monotherapy phase, all participants will receive vedolizumab intravenous infusion once at Weeks 30, 38, 46, 54, 62, 70, 78, 86, 94 and 102.

This multi-center trial will be conducted in the United States and Canada. The overall time to participate in this study is 128 weeks. Participants will make multiple visits to the clinic, plus a final visit 18 weeks after last dose of study drug for a safety follow-up assessment. Participants will also participate in a long-term safety questionnaire, by phone, at 26 weeks (6 months) from the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Has an initial diagnosis of CD established within 24 months prior to screening with involvement of the ileum and/or colon that can be assessed by ileocolonoscopy.
2. Has moderate to severely active CD during Screening defined by a centrally assessed simple endoscopic score for Crohn disease (SES-CD) score >=7 (or >=4 if isolated ileal disease).

Exclusion Criteria:

Gastrointestinal (GI) Exclusion Criteria

1. Has a diagnosis of ulcerative colitis (UC) or indeterminate colitis.
2. Has clinical evidence of a current abdominal abscess or a history of prior abdominal abscess.
3. Has a known perianal fistula with abscess. (The participant may have a perianal fistula without abscess.)
4. Has a known fistula (other than perianal fistula).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (32):
- United States (27):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Gastro Florida, Clearwater, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Northshore University HealthSystem, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cotton O'Neil Clinical Research, Topeka, Kansas
  - Texas Digestive Disease Consultants Baton Rouge, Baton Rouge, Louisiana
  - Louisana Research Center, LLC, Shreveport, Louisiana
  - Center for Digestive Health, Troy, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Minnesota Gastroenterology, PA - Plymouth, Plymouth, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Digestive Health Partners, PS, Asheville, North Carolina
  - Carolinas HealthCare System Digestive Health, Charlotte, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Baylor College of Medicine, Houston, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Texas Digestive Disease Consultants Southlake, Southlake, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Texas Digestive Disease Consultants, Webster, Webster, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Digestive Health Specialists, Tacoma, Washington
- Canada (5):
  - Covenant Health, Edmonton, Alberta
  - PerCuro Clinical Research Ltd, Victoria, British Columbia
  - LHSC - Victoria Hospital, London, Ontario
  - Toronto Digestive Disease Associates Inc, Vaughan, Ontario
  - CIUSSS de I'Estrie-CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Colombel JF, Ungaro RC, Sands BE, Siegel CA, Wolf DC, Valentine JF, Feagan BG, Neustifter B, Kadali H, Nazarey P, James A, Jairath V, Qasim Khan RM. Vedolizumab, Adalimumab, and Methotrexate Combination Therapy in Crohn's Disease (EXPLORER). Clin Gastroenterol Hepatol. 2024 Jul;22(7):1487-1496.e12. doi: 10.1016/j.cgh.2023.09.010. Epub 2023 Sep 22. PMID 37743037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in Canada and United States from 18 April 2017 to 05 July 2022.
Pre-assignment Details: Participants with newly-diagnosed Crohn's Disease (CD) with higher risk for complications were enrolled into triple combination therapy to assess efficacy and safety of vedolizumab 300 mg, adalimumab 160/80/40 mg, and methotrexate 15 mg, following monotherapy of vedolizumab 300 mg.
Groups:
- Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral): Participants received triple combination therapy of vedolizumab 300 milligram (mg), intravenous (IV) infusion, once at Weeks 0, 2, 6, 14 and 22, with adalimumab 160 mg subcutaneously (SC), once at Week 0, then 80 mg once at Week 2, then 40 mg once at Week 4 and every 2 weeks thereafter until Week 26 along with oral Methotrexate 15 mg tablets orally once weekly from Weeks 0 up to Week 34. Following the triple combination treatment participants received monotherapy of vedolizumab 300 mg IV infusion once at Weeks 30, 38, 46, 54, 62, 70, 78, 86, 94 and 102.
Period: Overall Study
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral)
Started | 55
Triple Combination Therapy (Participants who received triple combination therapy of vedolizumab 300 mg, IV infusion, adalimumab 160-80-40 mg SC and Methotrexate 15 mg tablets orally.) | 55
Monotherapy (Participants who received vedolizumab 300 mg IV infusion as monotherapy or have any visit data after Week 26 and before the safety follow up.) | 45
Safety Follow-up (Participants who completed the study treatment or were terminated early from the study were followed-up for safety up to 18 weeks after receiving the last dose of study drug.) | 53
Completed | 16
Not Completed | 39
Not completed — Pretreatment Event/Adverse Event | 9
Not completed — Lost to Follow-up | 4
Not completed — Voluntary Withdrawal | 8
Not completed — Site Termination | 1
Not completed — Lack of Efficacy | 16
Not completed — Reason not Specified | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15mg (Oral): Participants received triple combination therapy of vedolizumab 300 mg, IV infusion, once at Weeks 0, 2, 6, 14 and 22, with adalimumab 160 mg SC, once at Week 0, then 80 mg once at Week 2, then 40 mg once at Week 4 and every 2 weeks thereafter until Week 26 along with oral Methotrexate 15 mg tablets orally once weekly from Weeks 0 up to Week 34. Following the triple combination treatment participants received monotherapy of vedolizumab 300 mg IV infusion once at Weeks 30, 38, 46, 54, 62, 70, 78, 86, 94 and 102.
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15mg (Oral)
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 49
  More than one race | 1
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 171.4 (9.55)
Weight [Mean (Standard Deviation); unit: kg] | 71.87 (18.373)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated from the weight measured prior to the first dose of study drug and height taken at Screening. BMI=weight (kg)/height (m)^2.
  kg/m^2 | 24.26 (5.029)
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 14
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Endoscopic Remission at Week 26
Description: Endoscopic remission was defined as simple endoscopic score for Crohn's Disease (SES-CD) scale score from 0-2. The SES-CD evaluated 4 endoscopic variables: ulcer size, proportion of the surface area that was ulcerated, proportion of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable was the sum of values obtained for each segment. The SES-CD total was the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Week 26
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of study medication and have a post-enrollment efficacy assessment. As pre-specified in the protocol, this outcome measure reports data only in the Triple Combination Therapy Phase at Week 26.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral): Participants received triple combination therapy of vedolizumab 300 mg, IV infusion, once at Weeks 0, 2, 6, 14 and 22, with adalimumab 160 mg SC, once at Week 0, then 80 mg once at Week 2, then 40 mg once at Week 4 and every 2 weeks thereafter until Week 26 along with oral Methotrexate 15 mg tablets orally once weekly from Weeks 0 up to Week 34.
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral)
Number analyzed (Participants) | 55
percentage of participants | 34.5 [21.1 to 48.0]

2. Secondary Outcome: Percentage of Participants Achieving Endoscopic Healing at Week 26
Description: Endoscopic healing was defined as SES-CD score ≤4 and reduction from Baseline in SES-CD score of at least 2 points and no individual SES-CD subscore >1. The SES-CD evaluated 4 endoscopic variables: ulcer size, proportion of the surface area that is ulcerated, proportion of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable was the sum of values obtained for each segment. The SES-CD total was the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Percentages are rounded off to single decimal.
Time Frame: Week 26
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral)
Number analyzed (Participants) | 55
percentage of participants | 43.6 [29.6 to 57.7]

3. Secondary Outcome: Percentage of Participants Achieving Endoscopic Response at Week 26
Description: Endoscopic response was defined as 50% reduction in SES-CD score from Baseline. The SES-CD evaluated 4 endoscopic variables: ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable was sum of values obtained for each segment. The SES-CD total was the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Percentages are rounded off to single decimal.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral)
Number analyzed (Participants) | 55
percentage of participants | 56.4 [42.3 to 70.4]

4. Secondary Outcome: Change From Baseline in SES-CD Score at Week 26
Description: The SES-CD evaluated 4 endoscopic variables: ulcer size, proportion of the surface area that is ulcerated, proportion of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable was the sum of values obtained for each segment. The SES-CD total was the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Negative change indicates improvement.
Time Frame: Baseline and Week 26
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Number analyzed indicates the number of participants available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral)
Number analyzed (Participants) | 55
score on a scale
  Baseline | 12.6 (5.67)
  Change From Baseline at Week 26: number analyzed (Participants) | 45
  Change From Baseline at Week 26 | -8.9 (7.29)

5. Secondary Outcome: Percentage of Participants Achieving Deep Remission at Week 26
Description: Deep remission was defined as Crohn's disease activity index (CDAI) score <150 and SES-CD score from 0-2. CDAI was scoring system for the assessment of CD activity, index values of 150 and below were associated with quiescent disease; values above that indicated active disease and values above 450 were seen with extremely severe disease. The SES-CD evaluated 4 endoscopic variables: ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable was sum of values obtained for each segment. The SES-CD total was sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Percentages are rounded off to single decimal.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral)
Number analyzed (Participants) | 55
percentage of participants | 21.8 [10.0 to 33.6]

6. Secondary Outcome: Percentage of Participants Achieving Clinical Remission and Endoscopic Response as a Measure of Mucosal Healing at Week 26
Description: Clinical remission was defined as CDAI score <150. Endoscopic response was defined as 50% reduction in SES-CD score from Baseline, as mucosal healing. CDAI was scoring system for assessment of CD activity, index values of 150 and below are associated with quiescent disease; values above that indicated active disease and values above 450 were seen with extremely severe disease. The SES-CD evaluated 4 endoscopic variables: ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The SES-CD total was sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Percentages are rounded off to single decimal.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral)
Number analyzed (Participants) | 55
percentage of participants | 38.2 [24.4 to 51.9]

7. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Weeks 10 and 26
Description: Clinical remission was defined as CDAI score <150. CDAI was scoring system for the assessment of CD activity, index values of 150 and below were associated with quiescent disease; values above that indicated active disease and values above 450 were seen with extremely severe disease. Percentages are rounded off to single decimal.
Time Frame: Weeks 10 and 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral)
Number analyzed (Participants) | 55
percentage of participants
  Week 10 | 60.0 [46.1 to 73.9]
  Week 26 | 54.5 [40.5 to 68.6]

8. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Weeks 10 and 26
Description: Clinical response was defined as ≥100-point decrease in CDAI score. CDAI was scoring system for the assessment of CD activity, index values of 150 and below were associated with quiescent disease; values above that indicated active disease and values above 450 were seen with extremely severe disease. Percentages are rounded off to single decimal.
Time Frame: Weeks 10 and 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral)
Number analyzed (Participants) | 55
percentage of participants
  Week 10 | 49.1 [35.0 to 63.2]
  Week 26 | 43.6 [29.6 to 57.7]

9. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) Levels at Weeks 10 and 26
Description: The change between the CRP levels were collected at Weeks 10 and 26 relative to Baseline. Negative change indicates improvement.
Time Frame: Baseline, Weeks 10 and 26
Population: as for outcome 4
Measure: Median (Full Range); unit: milligrams per liter (mg/L)
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral)
Number analyzed (Participants) | 55
milligrams per liter (mg/L)
  Baseline | 7.60 [0.6 to 135.8]
  Change From Baseline at Week 10: number analyzed (Participants) | 49
  Change From Baseline at Week 10 | -4.80 [-84.0 to 29.7]
  Change From Baseline at Week 26: number analyzed (Participants) | 44
  Change From Baseline at Week 26 | -5.50 [-79.3 to 104.3]

10. Secondary Outcome: Change From Baseline in Fecal Calprotectin Concentrations at Weeks 10, 14, 26, 52, 78, and 102
Description: The change between the fecal calprotectin concentrations collected at Weeks 10, 14, 26, 52, 78, and 102 relative to Baseline were reported. Baseline is defined as the last observation prior to the first dose of the study drug.
Time Frame: Baseline, Weeks 10, 14, 26, 52, 78 and 102
Population: as for outcome 4
Measure: Median (Full Range); unit: micrograms per gram
Groups:
- Vedolizumab 300 mg (IV): Following the triple combination treatment participants received monotherapy of vedolizumab 300 mg IV infusion once at Weeks 30, 38, 46, 54, 62, 70, 78, 86, 94 and 102.
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral) | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 55 | 45
micrograms per gram
  Baseline | 1301.0 [23 to 17707] | 1210.0 [23 to 17707]
  Change From Baseline at Week 10: number analyzed (Participants) | 41 | 0
  Change From Baseline at Week 10 | -864.0 [-16406 to 471] |
  Change From Baseline at Week 14: number analyzed (Participants) | 44 | 0
  Change From Baseline at Week 14 | -556.0 [-14742 to 6892] |
  Change From Baseline at Week 26: number analyzed (Participants) | 36 | 0
  Change From Baseline at Week 26 | -860.5 [-7911 to 440] |
  Change From Baseline at Week 52: number analyzed (Participants) | 0 | 38
  Change From Baseline at Week 52 |  | -350.0 [-7365 to 8021]
  Change From Baseline at Week 78: number analyzed (Participants) | 0 | 26
  Change From Baseline at Week 78 |  | -396.5 [-7844 to 9434]
  Change From Baseline at Week 102: number analyzed (Participants) | 0 | 13
  Change From Baseline at Week 102 |  | -452.0 [-8052 to 106]

11. Secondary Outcome: Percentage of Participants Achieving Clinical Remission and CRP <5 Milligram Per Liter (mg/L) at Weeks 26, 52, 78, and 102
Description: Clinical remission was defined as CDAI score <150 and CRP level <5 mg/L in participants with elevated CRP level at Baseline. CDAI was scoring system for the assessment of CD activity, index values of 150 and below were associated with quiescent disease; values above that indicate active disease and values above 450 were seen with extremely severe disease. Percentages are rounded off to single decimal.
Time Frame: Weeks 26, 52, 78 and 102
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Overall number of participants analyzed are the number of participants with Elevated CRP at Baseline. Number analyzed indicates the number of participants available for analysis at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral) | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 39 | 34
percentage of participants
  Week 26: number analyzed (Participants) | 39 | 0
  Week 26 | 51.3 [34.3 to 68.3] |
  Week 52: number analyzed (Participants) | 0 | 34
  Week 52 |  | 44.1 [26.0 to 62.3]
  Week 78: number analyzed (Participants) | 0 | 34
  Week 78 |  | 26.5 [10.2 to 42.8]
  Week 102: number analyzed (Participants) | 0 | 34
  Week 102 |  | 20.6 [5.5 to 35.7]

12. Secondary Outcome: Percentage of Participants Using Oral Corticosteroids at Baseline Who Have Discontinued Corticosteroids and Are in Clinical Remission at Weeks 10, 26, and 102
Description: Percentage of participants using oral corticosteroids at Baseline who had discontinued corticosteroids and were in clinical remission at weeks 10, 26, and 102 were reported. Clinical remission was defined as CDAI score <150. CDAI was scoring system for the assessment of CD activity, index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 were seen with extremely severe disease. Percentages are rounded off to single decimal.
Time Frame: Weeks 10, 26 and 102
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Overall number of participants analyzed are the number of participants with Baseline concomitant oral corticosteroid use. Number analyzed indicates the number of participants available for analysis at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral) | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 16 | 14
percentage of participants
  Week 10: number analyzed (Participants) | 16 | 0
  Week 10 | 50.0 [22.4 to 77.6] |
  Week 26: number analyzed (Participants) | 16 | 0
  Week 26 | 56.3 [28.8 to 83.7] |
  Week 102: number analyzed (Participants) | 0 | 14
  Week 102 |  | 21.4 [0.0 to 46.5]

13. Secondary Outcome: Percentage of Participants Maintaining Clinical Remission at Weeks 52, 78, and 102
Description: Clinical remission was defined as CDAI score <150. Clinical remission was defined as CDAI score <150. CDAI was scoring system for the assessment of CD activity, index values of 150 and below are associated with quiescent disease; values above that indicated active disease and values above 450 were seen with extremely severe disease. Percentages are rounded off to single decimal.
Time Frame: Weeks 52, 78 and 102
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Overall number of participants analyzed are the number of participants with clinical remission at Week 26.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 30
percentage of participants
  Week 52 | 50.0 [30.4 to 69.6]
  Week 78 | 33.3 [14.8 to 51.9]
  Week 102 | 20.0 [4.0 to 36.0]

14. Secondary Outcome: Percentage of Participants Maintaining Clinical Response at Weeks 52, 78, and 102
Description: as for outcome 8
Time Frame: Weeks 52, 78 and 102
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Overall number of participants analyzed are the number of participants with clinical response at Week 26.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 24
percentage of participants
  Week 52 | 66.7 [45.7 to 87.6]
  Week 78 | 45.8 [23.8 to 67.9]
  Week 102 | 29.2 [8.9 to 49.4]

15. Secondary Outcome: Percentage of Participants Maintaining Endoscopic Remission at Week 102
Description: Endoscopic remission was defined as SES-CD score 0-2. The SES-CD evaluated 4 endoscopic variables: ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable was sum of values obtained for each segment. The SES-CD total was the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicated more severe disease. Percentages are rounded off to single decimal.
Time Frame: Week 102
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Overall number of participants analyzed are the number of participants with endoscopic remission at Week 26.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 18
percentage of participants | 27.8 [4.3 to 51.2]

16. Secondary Outcome: Percentage of Participants Maintaining Deep Remission at Week 102
Description: Deep remission was defined as CDAI score <150 and SES-CD score 0-2. Clinical remission was defined as CDAI score <150. CDAI was scoring system for the assessment of CD activity, index values of 150 and below are associated with quiescent disease; values above that indicated active disease and values above 450 were seen with extremely severe disease. The SES-CD evaluated 4 endoscopic variables: ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The SES-CD total was the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Percentages are rounded off to single decimal.
Time Frame: Week 102
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Overall number of participants analyzed are the number of participants with deep remission at Week 26.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 12
percentage of participants | 8.3 [0.0 to 28.1]

17. Secondary Outcome: Percentage of Participants Maintaining Endoscopic Healing at Week 102
Description: Endoscopic healing was defined as SES-CD score <=4 and reduction from Baseline in SES-CD score of at least 2 points and no individual SES-CD subscore >1. The SES-CD evaluated 4 endoscopic variables: ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable was sum of values obtained for each segment. The SES-CD total was the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Percentages are rounded off to single decimal.
Time Frame: Week 102
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Overall number of participants analyzed are the number of participants with endoscopic healing at Week 26.
Measure: Number (94% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 23
percentage of participants | 34.8 [13.1 to 56.4]

18. Secondary Outcome: Percentage of Participants Maintaining Endoscopic Response at Week 102
Description: Endoscopic response was defined as 50% reduction in SES-CD score from Baseline. The SES-CD evaluated 4 endoscopic variables: ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable was sum of values obtained for each segment. The SES-CD total was the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Week 102
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Overall number of participants analyzed are the number of participants with endoscopic response at Week 26.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 30
percentage of participants | 50.0 [30.4 to 69.6]

19. Secondary Outcome: Percentage of Participants Maintaining Clinical Remission and Endoscopic Response as a Measure of Mucosal Healing at Week 102
Description: Clinical remission is defined as CDAI score <150. Endoscopic response defined as 50% reduction in SES-CD score from Baseline, as mucosal healing. CDAI is scoring system for assessment of CD activity, index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease. The SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The SES-CD total is sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Percentages are rounded off to the nearest decimal value.
Time Frame: Week 102
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Overall number of participants analyzed are the number of participants with clinical remission and endoscopic response at Week 26.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 21
percentage of participants | 19.0 [0.0 to 38.2]

20. Secondary Outcome: Percentage of Participants With First Exacerbation of CD
Description: First exacerbation of CD after 26 weeks was defined as either: 1) a CDAI increase of >70 from the prior visit on 2 occasions separated by a 2-week interval, objective evidence of disease activity by colonoscopy or CRP above normal OR 2) fecal calprotectin >250 microgram per gram (mcg/g) alone. CDAI was scoring system for the assessment of CD activity, index values of 150 and below were associated with quiescent disease; values above that indicated active disease and values above 450 are seen with extremely severe disease. Percentages are rounded off to the nearest decimal value.
Time Frame: After 26 Weeks up to Week 120
Population: FAS included all participants who received at least 1 dose of study medication and had a post-enrollment efficacy assessment. Overall number of participants analyzed are the number of participants with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (IV)
Number analyzed (Participants) | 45
percentage of participants | 62.2 [46.9 to 77.5]

ADVERSE EVENTS:
Time Frame: From the first dose up to EOS (up to 120 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Data for the safety was collected and reported separately for triple combination therapy, monotherapy, and the safety follow up.
Groups:
- Safety Follow-up: Participants who completed the study treatment or were terminated early from the study were followed-up for safety up to 18 weeks after receiving the last dose of study drug.
Arm/Group | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral) | Vedolizumab 300 mg (IV) | Safety Follow-up
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/45 | 0/53
Serious Adverse Events (participants affected / at risk) | 6/55 | 1/45 | 2/53
Other Adverse Events (participants affected / at risk) | 36/55 | 31/45 | 4/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral) (N=55) | Vedolizumab 300 mg (IV) (N=45) | Safety Follow-up (N=53)
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (IV) + Adalimumab 160-80-40 mg (SC) + Methotrexate 15 mg (Oral) (N=55) | Vedolizumab 300 mg (IV) (N=45) | Safety Follow-up (N=53)
Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 2 | 0
C-reactive protein increased (Investigations) | 1 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Crohn's disease (Gastrointestinal disorders) | 9 | 20 | 4
Dizziness (Nervous system disorders) | 1 | 3 | 0
Faecal calprotectin increased (Investigations) | 2 | 4 | 0
Fatigue (General disorders) | 4 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 3 | 0
Headache (Nervous system disorders) | 5 | 2 | 0
Nasopharyngitis (Infections and infestations) | 6 | 3 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 0
Urinary tract infection (Infections and infestations) | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT02764762/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT02764762/SAP_002.pdf